CLINICAL TRIAL: NCT07186959
Title: A Novel Endoscopic Gastric Purse-string Suture Device for Weight Management in an in Vivo Human Model
Brief Title: EGPSS for Weight Management in an in Vivo Human Model
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Liu Yan (Other)
Responsible Party: Sponsor-Investigator, Liu Yan, Director, Head of Gastroenterology, Principal Investigator, Clinical Professor, Beijing 302 Hospital
Organization: Beijing 302 Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EGPSS for weight management
Record Dates: First submitted 2025-09-11; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Obesity, Mild
Keywords: obesity; endoscopic bariatric and metabolic therapy; bariatric surgery
MeSH Terms: conditions — Obesity; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Operation group (Experimental): Patients will undergo endoscopic gastric purse-string suturing procedure under endoscope by skilled endoscopist
  Interventions: Procedure: endoscopic gastric purse-string suturing

INTERVENTIONS:
Procedure: endoscopic gastric purse-string suturing — A dual-tail endoloop will be introduced into the stomach with endoscopic forceps, and will be secured to the gastric wall using endoscopic clips. An endoscope hook was used to tighten both tails of the endoloop until all the clips converged.

SUMMARY:
ndoscopic bariatric and metabolic therapies (EBMTs) have introduced more convenient, minimally invasive, and safe approaches to weight management. Mucosal ablation of the gastric fundus has been reported to limit fundic expansion and promote satiety; however, ablation can cause perforation, infection, bleeding, and other complications. To restrain fundic expansion while minimizing surgical trauma and preserving reversibility, an endoscopic gastric purse-string suturing (EGPSS) technique was developed to reduce gastric volume. This procedure may be suitable for short-term weight management. Safety and feasibility were demonstrated in a porcine model. The present study will evaluate the feasibility of EGPSS in participants with obesity and assess histological and physiological outcomes.

DETAILED DESCRIPTION:
The global prevalence of obesity has increased over the past five decades. Endoscopic bariatric and metabolic therapies (EBMTs) have introduced more convenient, minimally invasive, and safe approaches to weight management and have emerged as promising alternatives for treating obesity and related metabolic disorders (including type 2 diabetes and nonalcoholic fatty liver disease). Christopher et al. reported that ablation of the gastric fundus mucosa induces mucosal fibrosis; the resulting fibrotic tissue impedes fundic expansion and promotes satiety. However, fundic mucosal ablation may cause extensive and irreversible injury, increasing the risks of perforation, infection, bleeding, and other complications. A minimally invasive endoscopic therapy that inhibits fundic expansion while minimizing surgical trauma and preserving reversibility is therefore desirable.

Based on this rationale, an endoscopic gastric purse-string suturing (EGPSS) technique was developed to reduce the volume of the gastric fundus. EGPSS employs a specially designed endoclip in combination with an endoloop to appose the fundic mucosa and restrict fundic expansion. This procedure may be suitable for short-term weight management. Safety and feasibility have been demonstrated in a porcine model. The present study will evaluate the feasibility of EGPSS in participants with obesity and assess histological and physiological outcomes.

ELIGIBILITY:
Inclusion criteria:

* Patients with a body mass index (BMI) of 24-35 kg / m²;
* Patients accepted Lifestyle modifications, pharmacological interventions for weight loss which were unsuccessful or experienced a weight rebound;
* Patients willing to loss weight;
* Obese patients with metabolic disorders.

Exclusion criteria:

* Women who are planning to conceive, pregnant, or breastfeeding;
* Patients who are suffering from severe organ failure requiring hospitalization;
* Patients who have undergone gastrectomy;
* Patients allergic to anesthetics.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Percent Total Weight Loss (%TWL) measured by calibrated digital scale | Baseline and 3 months post-procedure
  Body weight recorded using a calibrated digital scale (kg). %TWL calculated as (baselineweight-follow-upweight)÷baselineweight × 100%. Measurements obtained under fasting conditions, light clothing, no shoes.

SECONDARY OUTCOMES:
Percent Excess Weight Loss (%EWL) measured by calibrated digital scale | Baseline and 3 months
  %EWL calculated as (baselineweight-follow-upweight)÷(baselineweight-idealweightatBMI25kg/m
  ) × 100%.
Satiety score (100-mm Visual Analog Scale, VAS) after standardized liquid meal | Baseline and 3 months
  Satiety assessed using a 100-mm VAS (0 = not at all, 100 = extremely) at 0, 15, 30, 60 minutes after a 400-kcal standardized liquid meal; area under the curve (AUC) computed.
Gastric fundus volume (magnetic resonance imaging, MRI) | Baseline and 3 months
  Fundic volume quantified by MRI volumetry during a standardized water-challenge protocol; primary read by a blinded radiologist; volume reported in mL and Δ from baseline.
Fasting plasma ghrelin and leptin (ELISA) | Baseline and 3 months
  Morning fasting venous samples analyzed by validated ELISA; concentrations reported in pg/mL (ghrelin) and ng/mL (leptin).
Insulin resistance (HOMA-IR) | Baseline and 3 months
  HOMA-IR calculated from fasting glucose (mmol/L) and insulin (µU/mL): insulin × glucose ÷ 22.5.
Procedure-related adverse events (ASGE lexicon severity grading) | Day 0 to Month 3
  All adverse events captured and coded using the ASGE lexicon with severity grade and relatedness adjudicated by the safety monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Liu, Principal Investigator — Beijing 302 Hospital
Locations (1):
- The fifth Medical Center of Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bluher M. Obesity: global epidemiology and pathogenesis. Nat Rev Endocrinol. 2019 May;15(5):288-298. doi: 10.1038/s41574-019-0176-8. PMID 30814686
- [Background] Maselli DB, Donnangelo LL, Coan B, McGowan CE. How to establish an endoscopic bariatric practice. World J Gastrointest Endosc. 2024 Apr 16;16(4):178-186. doi: 10.4253/wjge.v16.i4.178. PMID 38680199
- [Background] Simons M, Sharaiha RZ. Updates in metabolic bariatric endoscopy. Dig Endosc. 2024 Feb;36(2):107-115. doi: 10.1111/den.14633. Epub 2023 Aug 9. PMID 37405807
- [Background] Vargas EJ, Rizk M, Gomez-Villa J, Edwards PK, Jaruvongvanich V, Storm AC, Acosta A, Lake D, Fidler J, Bharucha AE, Camilleri M, Abu Dayyeh BK. Effect of endoscopic sleeve gastroplasty on gastric emptying, motility and hormones: a comparative prospective study. Gut. 2023 Jun;72(6):1073-1080. doi: 10.1136/gutjnl-2022-327816. Epub 2022 Oct 14. PMID 36241388